CLINICAL TRIAL: NCT00275431
Title: A Phase II, Open Label, Multicenter Study of Single-Agent AT-101 in Patients With Relapsed or Refractory B-Cell Malignancies (Follicular Lymphoma, Mantle Cell Lymphoma, Diffuse Large Cell Lymphoma, or Small Lymphocytic Lymphoma/Chronic Lymphocytic Leukemia)
Brief Title: Phase II Safety and Efficacy Study of Single-agent AT-101 in Patients With Relapsed or Refractory B-cell Malignancies
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ascenta Therapeutics (Industry)
Responsible Party: Lance Leopold, Ascenta Therapeutics, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AT-101-CS-005
Record Dates: First submitted 2006-01-10; First posted 2006-01-12 (Estimated); Last update posted 2011-06-29 (Estimated); Status verified 2011-06

CONDITIONS: Follicular Lymphoma; Diffuse Large Cell Lymphoma; Mantle Cell Lymphoma; Small Lymphocytic Lymphoma; Chronic Lymphocytic Leukemia
Keywords: cancer; AT-101; AT101; B-cell malignancies; Non-Hodgkin; lymphoma; lukemia
MeSH Terms: conditions — Lymphoma, Follicular; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Mantle-Cell; Leukemia, Lymphocytic, Chronic, B-Cell; Neoplasms; Lymphoma | interventions — gossypol acetic acid

INTERVENTIONS:
Drug: AT-101 — Oral

SUMMARY:
This is an open-label, multicenter, phase II study to evaluate the safety and efficacy of single-agent AT-101 in patients with relapsed or refractory B-cell malignancies.

DETAILED DESCRIPTION:
This is an open-label, multicenter, phase II study to evaluate the safety and efficacy of single-agent AT-101 in patients with relapsed or refractory B-cell malignancies. For the purpose of this study, B-cell malignancies can include one of the following disease sub-types: follicular lymphoma (FL), diffuse large b-cell lymphoma (DLBCL), mantle cell lymphoma (MCL), small lymphocytic lymphoma (SLL)/chronic lymphocytic leukemia. Patients will be enrolled according to disease subtype into one of four groups in two stages. The first stage of each group will enrolled 13 patients. If patients within any group experience disease response, an additional 14 patients will be enrolled into that group.

ELIGIBILITY:
Inclusion Criteria:

* Must have a histologically confirmed B-cell malignancy (defined as FL [any grade], DLBCL, MCL or SLL/CLL);
* Male or non-pregnant, non-lactating females age ≥18 years;
* Ability to swallow and retain oral medication.;
* Have failed at least one prior therapy and have documentation of either, relapsed disease, or refractory disease (i.e., no response or stable disease on their last regimen of therapy);
* ECOG performance status 0 or 1;
* All clinically significant toxicities from prior therapy must have fully resolved;
* Must have discontinued treatment with monoclonal antibodies for a minimum of 90 days prior to first dose of AT-101, or have objective documentation of disease progression if within 90 days of monoclonal antibody administration;
* Patients with FL, DLBCL, MCL, and SLL with normal lymphocyte counts must have at least one bi-dimensional lesion that is radiographically measurable (skin lesions, palpable lymph nodes, and bone marrow as the only site of disease are not considered measurable disease);
* Patients with SLL whose lymphocytes are elevated at baseline or CLL must have palpable lymph nodes and/or disease localized to the bone marrow per the NCI-Sponsored Working Group Guidelines for CLL.

Exclusion Criteria:

* Requirement of systemic corticosteroids within 7 days prior to and during AT-101 administration;
* Must not have received anti-cancer therapy within 28 days of first dose of AT-101. Cannot have received hormonal agents or biologic dose modifiers (with the exception of HRT) or any investigational treatments within 28 days of treatment with AT-101;
* Patients with CNS lymphoma, HIV-related lymphoma, symptoms suggesting HIV infection or active auto-immune hemolytic anemia are excluded;
* Previous treatment with gossypol, or are hypersensitive to its excipient are excluded;
* Patients who have an uncontrolled, concurrent illness are also excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2005-11; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Complete or partial remission of disease. | every 6 weeks

SECONDARY OUTCOMES:
Number of participants with adverse events. | every 3 weeks
duration of response | every 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Lance Leopold, MD, Study Director — Ascenta Therapeutics, Inc.
Locations (11):
- United States (11):
  - Birmingham, Alabama
  - San Diego, California
  - Atlanta, Georgia
  - Chicago, Illinois
  - Boston, Massachusetts
  - New York, New York
  - Rochester, New York
  - High Point, North Carolina
  - Hilton Head Island, South Carolina
  - Memphis, Tennessee
  - Burlington, Vermont